CLINICAL TRIAL: NCT06511505
Title: NOrthwestern Tempus AI-enaBLed Electrocardiography (NOTABLE) Trial: A Pragmatic, Real-world Study of an Artificial-intelligence Enabled Electrocardiogram Algorithms to Improve the Diagnosis of Cardiovascular Disease
Brief Title: NOrthwestern Tempus AI-enaBLed Electrocardiography (NOTABLE) Trial
Acronym: NOTABLE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Sanjiv Shah, Director, Institute for Artificial Intelligence in Medicine - Center for Deep Phenotyping and Precision Therapeutics, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STU00220862
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Atrial Fibrillation; Cardiovascular Diseases; Arrhythmia; Valvular Disease
Keywords: early detection; artificial intelligence; structural heart disease; atrial fibrillation; cardiac diagnostics
MeSH Terms: conditions — Atrial Fibrillation; Cardiovascular Diseases; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention (Experimental): Care teams randomized to the intervention will have access to the AI-enabled ECG-based screening tool.
  Interventions: Other: TEMPUS AI-enabled ECG-based Screening Tool
- Control (No Intervention): Care teams randomized to control will continue routine practice without access to the AI-enabled ECG-based screening tool.

INTERVENTIONS:
Other: TEMPUS AI-enabled ECG-based Screening Tool — The AI-enabled ECG-based screening tool, Tempus Next software, analyzes 12-lead ECG recordings to identify patients at increased risk for undiagnosed cardiovascular diseases, specifically atrial fibrillation (AF) and structural heart disease (SHD). Clinicians in the intervention group will receive a risk assessment for AF and SHD each time they order an ECG for their patients.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to determine if a machine learning/artificial intelligence (AI)-based electrocardiogram (ECG) algorithm (Tempus Next software) can identify undiagnosed cardiovascular disease in patients. It will also examine the safety and effectiveness of using this AI-based tool in a clinical setting. The main questions it aims to answer are:

1. Can the AI-based ECG algorithm improve the detection of atrial fibrillation and structural heart disease?
2. How does the use of this algorithm affect clinical decision-making and patient outcomes? Researchers will compare the outcomes of healthcare providers who receive the AI-based ECG results to those who do not.

Participants (healthcare providers) will:

Be randomized into two groups: one that receives AI-based ECG results and one that does not.

In the intervention group, receive an assessment of their patient's risk of atrial fibrillation or structural heart disease with each ordered ECG.

Decide whether to perform further clinical evaluation based on the AI-generated risk assessment as part of routine clinical care.

DETAILED DESCRIPTION:
There is a large burden of undiagnosed, treatable cardiovascular disease (CVD), encompassing various heart conditions such as arrhythmias (e.g., atrial fibrillation) and structural heart diseases (e.g., valvular disease). Early detection and accurate diagnosis can significantly improve patient outcomes by enabling timely, guideline-based interventions or therapies.

The goal of this study is to leverage machine learning approaches to enhance the detection and diagnosis of CVD. By identifying patients at risk of undiagnosed CVD and referring them for further clinical evaluation, we aim to improve health outcomes.

Study Overview:

The NOTABLE study will compare the rates of new disease diagnoses, therapeutic interventions, and cardiovascular outcomes between two groups of patients managed by clinicians at Northwestern Medicine:

Patients whose clinicians use ECG predictive models. Patients whose clinicians do not use ECG predictive models.

Intervention Details:

This study utilizes the Tempus Next software, which includes AI algorithms for analyzing 12-lead ECGs. Clinicians randomized to the intervention group will automatically receive an ECG with "Risk-Based Assessment for Cardiac Dysfunction" when ordering a 12-lead ECG within EPIC during the study period. If a high-risk result is identified, clinicians will receive an EHR inbox message recommending a follow-up diagnostic test, such as echocardiography and/or ambulatory ECG monitoring.

Outcome Tracking:

A monthly report will track and provide data on:

The proportion of patients with a high-risk result. The proportion of patients receiving the follow-up diagnostic test. The proportion of patients receiving guideline-recommended therapies. This report will be sent to the study participants and clinicians randomized to the intervention group. Clinicians in the usual care group will not receive any communication from the study investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Atrial fibrillation algorithm

   1. Age 65 or over
   2. ECG obtained as part of routine clinical care
2. Structural heart disease algorithm

   1. Age 40 or over
   2. ECG obtained as part of routine clinical care

Exclusion Criteria:

1. Atrial fibrillation algorithm

   1. No history of AF
   2. No permanent pacemaker (PPM) or implantable cardioverter defibrillator (ICD)
   3. No recent cardiac surgery (within the preceding 30 days)
2. Structural heart disease algorithm

   1. No history of SHD
   2. No echocardiogram within the past 1 year

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-08-03 (Estimated); Primary Completion 2025-08-03 (Estimated); Study Completion 2026-02-03 (Estimated)

PRIMARY OUTCOMES:
Rate of new CV diagnoses at 6 months | 6 months
  Rate of new CV diagnoses will be defined for each predictive model and a composite of all models, and comparisons will be made between intervention and control groups.
  AF: New AF diagnosis SHD: New diagnosis of moderate or severe aortic stenosis, aortic regurgitation, or mitral stenosis, new diagnosis of severe mitral regurgitation or tricuspid regurgitation, new diagnosis of LVEF ≤40%, new diagnosis of significant left ventricular hypertrophy (IVSd >15 mm).

SECONDARY OUTCOMES:
Rate of new CV therapies at 6 months | 6 months
  Rate of new CV therapies will be evaluated for each predictive model and a composite of all models, comparisons will be made between intervention and control groups.
  AF: antiarrhythmic use, AV nodal blocking agent use, anticoagulation use, AF ablation procedure SHD: new use of medication for LV systolic dysfunction (beta blockers, ACE-I/ARB/ARNI, MRA, SGLT2-I), new therapies for valvular heart disease (valve repair or replacement), new therapies for HCM, cardiac amyloidosis, hypertensive heart disease.
Rate of CV outcomes at 6 months | 6 months
  Rate of CV outcomes including CV death, MI, and hospitalization for a cardiovascular cause (including heart failure and stroke) between intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Shah, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States